CLINICAL TRIAL: NCT04155697
Title: Thirdhand Smoke Contamination in a Neonatal Intensive Care Unit (NICU)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thomas Francis Northrup, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-15-0614 (sub-study); R03HD088847 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Nicotine Exposure
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hand washing with soap for thirdhand smoke removal (Active Comparator)
  Interventions: Drug: 2% Chlorohexidine Gluconate soap
- Ethyl alcohol-based sanitizer for thirdhand smoke removal (Active Comparator)
  Interventions: Drug: 62% ethyl alcohol-based hand sanitizer

INTERVENTIONS:
Drug: 2% Chlorohexidine Gluconate soap — Participants will wash hands for 30 seconds with 2% Chlorohexidine Gluconate soap.
  Arms: Hand washing with soap for thirdhand smoke removal
Drug: 62% ethyl alcohol-based hand sanitizer — Participants will apply 62% ethyl alcohol-based hand sanitizer for 30 seconds
  Arms: Ethyl alcohol-based sanitizer for thirdhand smoke removal

SUMMARY:
The purpose of the study is to quantify the efficacy of hand washing (HW) and ethyl alcohol-based hand sanitizer (S) for third-hand smoke (THS) removal in a sub-sample of non-staff smokers using nicotine wipes on adjacent fingers before and after HW/S.

The hypotheses are that detectable levels of surface nicotine will remain on participants' fingers, regardless of hand washing (HW) and ethyl alcohol-based hand sanitizer (S) attempts and that greater finger levels of surface nicotine will remain after alcohol sanitization compared to hand washing.

ELIGIBILITY:
Inclusion Criteria ():

* Any non-staff participants visiting the NICU (including friends and family members of the infants' caregivers)
* Consented to and provided a finger wipe
* Report being a smoker
* Smoking status verified by an exhaled carbon monoxide (CO) level of >7 parts per million

Exclusion Criteria:

* Unwilling to comply with research procedures (i.e., finger wipes)
* Does not speak English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Nicotine level on finger #1 | baseline
  Nicotine will be sampled from one finger of each participant's dominant hand (thumb, index, or middle finger). Finger will be wiped and nicotine level will be quantified.
Nicotine level on finger #2 | 5 minutes after hand washing or sanitizing
  Nicotine will be sampled from one finger of each participant's dominant hand (thumb, index, or middle finger). Finger will be wiped and nicotine level will be quantified.
Nicotine level on finger #3 | 1 hour after hand washing or sanitizing
  Nicotine will be sampled from one finger of each participant's dominant hand (thumb, index, or middle finger). Finger will be wiped and nicotine level will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Northrup, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Northrup TF, Stotts AL, Suchting R, Khan AM, Klawans MR, Green C, Hoh E, Hovell MF, Matt GE, Quintana PJE. Handwashing Results in Incomplete Nicotine Removal from Fingers of Individuals who Smoke: A Randomized Controlled Experiment. Am J Perinatol. 2022 Nov;39(15):1634-1642. doi: 10.1055/s-0041-1736287. Epub 2021 Oct 11. PMID 34634832

DOCUMENTS (1):
  • Informed Consent Form (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04155697/ICF_000.pdf